CLINICAL TRIAL: NCT06058156
Title: A Multinational, Multicenter, Double-blind, Placebo-controlled Phase 2 Study to Evaluate Efficacy and Safety of SAR444656 in Adult Participants With Moderate to Severe Atopic Dermatitis
Brief Title: Phase 2 Study of SAR444656 in Adult Participants With Moderate to Severe Atopic Dermatitis
Acronym: ADVANTA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision. Not related to safety concern.
Sponsor: Sanofi (Industry)
Collaborators: Kymera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT17754; 2023-504346-66 (Registry Identifier: CTIS); U1111-1287-6919 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAR444656 dose 1 (Experimental): Participants will receive SAR444656 dose 1 orally
  Interventions: Drug: SAR444656 (KT-474)
- SAR444656 dose 2 (Experimental): Participants will receive SAR444656 dose 2 orally
  Interventions: Drug: SAR444656 (KT-474)
- SAR444656 dose 3 (Experimental): Participants will receive SAR444656 dose 3 orally
  Interventions: Drug: SAR444656 (KT-474)
- Placebo (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR444656 (KT-474) — Oral Tablet
  Arms: SAR444656 dose 1; SAR444656 dose 2; SAR444656 dose 3
Drug: Placebo — Oral Tablet
  Arms: Placebo

SUMMARY:
This is a multinational, multicenter, double-blind, placebo-controlled, parallel-group Phase 2, 4-arm study in adult participants with moderate to severe AD who are inadequately controlled with topical therapies or for whom such topical therapies are inadvisable and who are candidates for systemic therapy.

Participants will be randomized to receive SAR444656 dose 1, dose 2, dose 3 or matching placebo.

Participants who meet inclusion/exclusion criteria will be stratified for randomization by severity of AD (moderate [baseline EASI score <22] versus severe [baseline EASI score ≥22]).

The total duration of study is approximately 24 weeks, including 1 to 4 weeks for screening, 16 weeks for double-blind study treatment and 4 weeks for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants with atopic dermatitis as defined by the American Academy of Dermatology Consensus Criteria for at least 1 year before the baseline visit.
* EASI ≥12 at screening and at baseline visit
* vIGA score ≥3 (on the 0 to 4 IGA scale, in which 3 is moderate and 4 is severe) at screening and baseline visit.
* AD involvement ≥10% of BSA at screening and baseline visit
* Baseline PP-NRS ≥4
* Participants must have documented history within 6 months prior to baseline visit, of either inadequate response or inadvisability to topical medications
* Participants must have applied daily topical emollient (moisturizer) for at least the 7 consecutive days immediately before the baseline visit. Participants should continue using daily moisturizers during the study.
* Participants must be willing and able to complete the electronic diary for the duration of the study as required by the study protocol.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Presence of other skin conditions that may interfere with study assessments such as psoriasis, tinea corporis, lupus erythematosus
* Any active or chronic infection requiring systemic treatment within 4 weeks prior to baseline
* Known history of, or suspected, significant current immunosuppression, including history of invasive opportunistic or helminth infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration.
* History of solid organ or stem cell transplant.
* Participants with history of splenectomy.
* Participants with history of any malignancy or lymphoproliferative disease, except if the participant has been free from disease for ≥5 years. Successfully treated non-metastatic cutaneous squamous cell carcinoma, basal cell carcinoma, or localized carcinoma in situ of the cervix are allowed.
* Family history of sudden death or long QT syndrome.
* History of congenital or drug-induced long QT syndrome.
* Congestive heart failure (NYHA Class 2-4), greater than Class 1 angina pectoris, acute coronary syndrome within prior 6 months, known structural heart disease.
* History of any major cardiovascular events (eg, myocardial infarction, unstable angina pectoris, coronary revascularization, stroke, or transient ischemic attack) at any time prior to screening.
* History of ventricular fibrillation, ventricular tachycardia, Torsades de Pointes, atrial fibrillation, syncope not explained by non-cardiac etiology.
* Uncontrolled hypertension defined as consistent systolic blood pressure ≥150 mm Hg or consistent diastolic blood pressure ≥90 mm Hg despite antihypertensive medication.
* Participants had major surgery within 4 weeks prior to the screening or have planned any elective major surgery during the study.
* Having received any of protocol-specified prohibited therapy (Topical or systemic) within the specified timeframe prior to the baseline visit.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in EASI | Week 16
  Eczema area severity index is an Investigator-assessed validated tool used to measure the extent (area) and severity of atopic dermatitis (AD). Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.

SECONDARY OUTCOMES:
Proportion of participants with validated Investigational Global Assessment (vIGA)-AD of 0 or 1 and a reduction from baseline of ≥2 points | Week 16
Proportion of participants achieving EASI-75 (reduction of EASI score by ≥75% from baseline) | Week 16
Absolute change from baseline in EASI | Week 16
Proportion of participants achieving EASI-50 (reduction of EASI score by ≥50% from baseline) | Week 16
Proportion of participants achieving EASI-90 (reduction of EASI score by ≥90% from baseline) | Week 16
Change from baseline in percent body surface area (BSA) affected by AD | Week 16
Proportion of participants with reduction of weekly average of daily peak pruritus numeric rating scale (PP-NRS) by ≥4 points from baseline | Week 16
Percent change from baseline in weekly average of daily PP-NRS | Week 16
Absolute change from baseline in weekly average of daily PP-NRS | Week 16
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and adverse events of special interest (AESIs), investigational medicinal product (IMP) discontinuation due to TEAEs | Up to Week 20
Plasma SAR444656 concentration | Week 0, Week 1, Week 2, Week 4, and Week 16

CONTACTS AND LOCATIONS:
Locations (37):
- United States (10):
  - Clear Dermatology & Aesthetics Center- Site Number : 8400003, Scottsdale, Arizona
  - Encore Medical Research of Boynton Beach- Site Number : 8400002, Boynton Beach, Florida
  - Revival Research - Doral- Site Number : 8400007, Doral, Florida
  - Encore Medical Research - 6600 Taft St- Site Number : 8400004, Hollywood, Florida
  - Sullivan Dermatology- Site Number : 8400001, Miami, Florida
  - ARA Professionals- Site Number : 8400017, Miami, Florida
  - Encore Medical Research - Weston- Site Number : 8400008, Weston, Florida
  - Wayne Health - Dearborn- Site Number : 8400009, Dearborn, Michigan
  - UPMC Montefiore- Site Number : 8400006, Pittsburgh, Pennsylvania
  - ACRC Trials - Carrollton - Hunt - PPDS- Site Number : 8400012, Carrollton, Texas
- Czechia (3):
  - Investigational Site Number : 2030002, Ostrava
  - Investigational Site Number : 2030001, Pardubice
  - Investigational Site Number : 2030003, Prague
- Germany (8):
  - Investigational Site Number : 2760007, Heidelberg, Baden-Wurttemberg
  - Investigational Site Number : 2760009, Munich, Bavaria
  - Investigational Site Number : 2760008, Frankfurt am Main, Hesse
  - Investigational Site Number : 2760002, Buxtehude, Lower Saxony
  - Investigational Site Number : 2760003, Bochum, North Rhine-Westphalia
  - Investigational Site Number : 2760006, Remscheid, North Rhine-Westphalia
  - Investigational Site Number : 2760010, Dessau, Saxony-Anhalt
  - Investigational Site Number : 2760001, Berlin
- Greece (2):
  - Investigational Site Number : 3000001, Pavlos Melas, Thessaloniki
  - Investigational Site Number : 3000002, Thessaloniki
- Poland (11):
  - Investigational Site Number : 6160006, Tarnów, Lesser Poland Voivodeship
  - Investigational Site Number : 6160012, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160002, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160011, Lodz, Lódzkie
  - Investigational Site Number : 6160001, Lodz, Lódzkie
  - Investigational Site Number : 6160007, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160005, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160003, Chojnice, Pomeranian Voivodeship
  - Investigational Site Number : 6160004, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6160009, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160010, Lodz
- South Korea (3):
  - Investigational Site Number : 4100002, Cheonan-si, Chungcheongnam-do
  - Investigational Site Number : 4100001, Ansan-si, Gyeonggi-do
  - Investigational Site Number : 4100004, Seongbuk-Gu, Seoul-teukbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT17754 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25557&tenant=MT_SNY_9011